CLINICAL TRIAL: NCT00881387
Title: A Pilot Study of Rituximab-Gemcitabine-Navelbine for Relapsed/Refractory Hodgkin's Lymphoma
Brief Title: Rituximab, Gemcitabine, and Vinorelbine in Treating Patients With Hodgkin Lymphoma That Has Relapsed or Not Responded to Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080919; SCCC-2007092
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Rituximab; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (eligible for SCT) (Experimental): Patients receive rituximab IV, vinorelbine ditartrate IV over 6-10 minutes, and gemcitabine hydrochloride IV over 30 minutes on day 1 and pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) or partial response (PR) undergo SCT.
  Interventions: Biological: rituximab; Drug: gemcitabine hydrochloride; Drug: vinorelbine ditartrate
- Group 2 (ineligible for SCT) (Experimental): Patients receive rituximab, vinorelbine ditartrate, gemcitabine hydrochloride, and pegfilgrastim as in group 1. Patients with CR, PR, or stable disease after 3 courses continue to receive therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: gemcitabine hydrochloride; Drug: vinorelbine ditartrate

INTERVENTIONS:
Biological: rituximab — Given IV
Drug: gemcitabine hydrochloride — Given IV
Drug: vinorelbine ditartrate — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Drugs used in chemotherapy, such as gemcitabine and vinorelbine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with gemcitabine and vinorelbine may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with gemcitabine and vinorelbine works in treating patients with Hodgkin lymphoma that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the response rate (complete response/remission, unconfirmed complete response, partial response/remission) in patients with relapsed or refractory Hodgkin lymphoma treated with 3 courses of rituximab, gemcitabine hydrochloride, and vinorelbine ditartrate.

Secondary

* Assess progression-free survival, failure-free survival, and overall survival of patients treated with this regimen.
* Characterize the safety profile of this regimen in these patients.
* Determine the rate of adequate stem cell collection (≥ 2 million CD34+ cells) in patients eligible for stem cell transplantation.

OUTLINE: Patients are assigned to 1 of 2 treatment groups according to eligibility for stem cell transplantation (SCT).

* Group 1 (eligible for SCT): Patients receive rituximab IV, vinorelbine ditartrate IV over 6-10 minutes, and gemcitabine hydrochloride IV over 30 minutes on day 1 and pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) or partial response (PR) undergo SCT.
* Group 2 (ineligible for SCT): Patients receive rituximab, vinorelbine ditartrate, gemcitabine hydrochloride, and pegfilgrastim as in group 1. Patients with CR, PR, or stable disease after 3 courses continue to receive therapy in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed for at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed classical Hodgkin lymphoma, including 1 of the following cell types:

  * Nodular sclerosis
  * Mixed cellularity
  * Lymphocyte-rich
  * Lymphocyte-depleted
* Measurable disease using the Cheson criteria, defined as ≥ 1 unidimensionally measurable lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* Progressive or relapsed disease after ≥ 1 prior line of combination chemotherapy
* No known CNS metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC > 1,500/mm^3
* Platelet count > 75,000/mm^3
* Total bilirubin ≤ 2 mg/dL (unless due to hemolysis)
* AST or ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active hepatitis B infection
* No known chronic hepatitis B carrier
* No HIV positivity
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Symptomatic neurological illness
  * Active uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant at the time of study treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Significant pulmonary disease or hypoxia
  * Psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 14 days since prior chemotherapy, immunotherapy, biological therapy, or investigational therapy and recovered
* No prior gemcitabine hydrochloride, vinorelbine ditartrate, or rituximab
* No other concurrent investigational or commercial agents or therapies with the intent to treat the malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response, unconfirmed complete response, partial response) | After first 3 cycles of treatment

SECONDARY OUTCOMES:
Progression-free survival, failure-free survival, and overall survival | Treatment start date to date of death for any reason
Safety profile | Cycle 1 Day 1 through Follow-up
Rate of adequate stem cell collection | After completion of 3 cycle of treatment
  This will be assessed only for patients eligible for stem-cell transplantation after completion of R-Gemzar/Navelbine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Stefanovic, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States